CLINICAL TRIAL: NCT03562767
Title: A Randomized Single Blinded Interventional Study to Assess the Feasibility and Acceptability of a Culturally-Tailored Cognitive Behavior Intervention (CT-CB) for African American Patients With Uncontrolled Type 2 Diabetes and to Compare the Effects of Intervention to Standard of Care on Diabetes Control Measures.
Brief Title: Cognitive Behavioral Therapy for African Americans With Uncontrolled Type-2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A control group was intended to be added to the study, but the study team decided not complete this additional research with the pandemic. Additional funds were also not available to enroll a new control group and thus, the study was terminated.
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ambar Kulshreshtha, Assistant Professor, Department of Family and Preventive Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00101847; P30DK111024 (NIH)
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Results first posted 2022-01-03 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Culturally-Tailored Cognitive Behavior intervention (CT-CB); Family Practice; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Three groups of subjects with uncontrolled diabetes Type 2 will be followed longitudinally for 3 months
Who Masked: Outcomes Assessor
Masking Description: Research staff conducting the psychological, physical, outcome assessments, and study analyses will be blinded to participant's group allocation. To minimize bias, participants in the intervention group will be asked to refrain from disclosing their group assignment to study staff who collect data and questionnaires. Due to the overt nature of the CT-CB approach, the investigators and participants in the intervention group will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-based Cognitive Behavioral Intervention (Experimental): Subjects receiving the group-based CT-CB intervention
  Interventions: Behavioral: Group-based Cognitive Behavioral Intervention
- Web-based Cognitive Behavioral Intervention (Experimental): Subjects receiving the web based CT-CB intervention
  Interventions: Behavioral: Web-based Cognitive Behavioral Intervention
- Usual Care (Placebo Comparator): Subjects receiving usual care from their primary care providers
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Group-based Cognitive Behavioral Intervention — This intervention will include six 1-hour group sessions held biweekly for twelve weeks. Each sixty-minute session will consist of 15 minutes of diabetes education regarding exercise and food planning and approximately 45 minutes of CT-CB presentations/engagement activities. Participants will be encouraged to bring along their family members or friends for support.
  Arms: Group-based Cognitive Behavioral Intervention
Behavioral: Web-based Cognitive Behavioral Intervention — This intervention will include six 1-hour web-based sessions held biweekly for twelve weeks. Subjects in the web-based CT-CB will be asked to reserve a 1 hour period for a web call from the Behavioral Interventionist team. Text reminders will be sent to the participants prior the sessions. During this period, approximately 15 minutes will be reserved for diabetes exercise and food planning education and approximately 45 minutes of CT-CB engagement activities.
  Arms: Web-based Cognitive Behavioral Intervention
Behavioral: Usual Care — Usual care group participants will continue to receive care and follow up from their primary care providers as per the American Diabetes Association guidelines with log books, education regarding self-management strategies and appropriate referrals as needed.
  Arms: Usual Care

SUMMARY:
The main purpose of the study is to assess the feasibility and acceptability of a Culturally-Tailored Cognitive Behavior intervention (CT-CB) for African American patients with uncontrolled Type 2 diabetes. After the baseline visit subjects will be randomly assigned to undergo a six session group-based or web-based behavioral intervention (CT-CB) program or to general education (usual care). The intervention duration is 12 weeks.

DETAILED DESCRIPTION:
African Americans are approximately twice as likely to be diagnosed with diabetes and to experience gaps in diabetes care compared to Whites. Lower health literacy and socio-economic, language, and communication barriers are all associated with disparities in diabetes care. The role of Behavioral theory is foundational in understanding behavior change among patients in the self-management of diabetes. Further culturally tailoring increases acceptance and effectiveness of diabetes self-management.

The aim of this pilot study is to test the feasibility and acceptability of a culturally tailored, cognitive behavioral intervention (CT-CB) program using a group-based vs. a web-based format, and determine if it can improve diabetes self-management among African Americans compared with usual individual based care at the clinic. Forty-five African American patients with uncontrolled type 2 diabetes (HbA1C > 8 %), aged > 18 years, will be randomly assigned to undergo a six session group-based or web-based behavioral intervention (CT-CB) program or to general education (usual care). After 12 weeks, patients will be followed for an additional three months to evaluate for diminution of treatment effects. Both the group -based and the web-based CBT intervention group will be followed for an additional three months to study for possible diminution of treatment effects over time.

Diabetic measures like Hemoglobin (HbA1C) at baseline vs. 3 months; the Patient Health Questionnaire to assess depressive symptoms; Diabetes Distress Scale, anxiety, self-efficacy, quality of life (SF-12), Diabetes Health Belief Scale, process measures such as Patient Activation Measure (PAM-13), medication adherence questionnaire, session-participation, glucose self-monitoring, diet and physical activity are measured at each visit pre and post intervention. Trained study staff will also conduct neuropsychological tests including language and memory tests, attention and executive function tests, clinical diagnosis, activities of daily living (ADL).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Fluency in English
* African American
* HbA1C>8%

Exclusion Criteria:

* Subjects with no web access,
* Subjects using an insulin pump,
* Subjects that are pregnant
* Subjects that have active substance abuse including alcohol,
* Subjects with visual impairment or have severe hearing or other physical disabilities that would be a barrier for participating in-group or web sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ambar Kulshreshtha, MD, PhD FAHA, Principal Investigator — Emory University
Locations (1):
- Emory Dunwoody Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share the participants data

REFERENCES:
- [Derived] Cornely RM, Subramanya V, Owen A, McGee RE, Kulshreshtha A. A mixed-methods approach to understanding the perspectives, experiences, and attitudes of a culturally tailored cognitive behavioral therapy/motivational interviewing intervention for African American patients with type 2 diabetes: a randomized parallel design pilot study. Pilot Feasibility Stud. 2022 May 21;8(1):107. doi: 10.1186/s40814-022-01066-4. PMID 35597972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A control group was intended to be added to the study, but the study team decided not to complete this additional research due to the pandemic. Additional funds were not available to enroll a new control group and thus, the study was terminated.
Period: Overall Study
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention | Usual Care
Started | 10 | 10 | 0
Completed | 7 | 7 | 0
Not Completed | 3 | 3 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Logistic Reason | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: A control group was intended to be added to the study, but the study team decided not to complete this additional research due to the pandemic. Additional funds were not available to enroll a new control group and thus, the study was terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention | Usual Care | Total
Number analyzed (Participants) | 7 | 7 | 0 | 14
Age, Customized [Count of Participants; unit: Participants]
  <55 Years Old | 4 | 1 | 0 | 5
  ≥55 Years Old | 3 | 6 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 |  | 11
  Male | 2 | 1 |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 0 | 14
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 |  | 14
BMI [Count of Participants; unit: Participants]
  Normal (BMI 18.5-24.9 kg/m^2) | 1 | 1 | 0 | 2
  Overweight (BMI 25.0-29.9 kg/m^2) | 1 | 2 | 0 | 3
  Obese (BMI >= 30.0 kg/m^2) | 5 | 4 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Complete the Study Compared to Enrolled
Description: Feasibility of the intervention will be measured as the percentage of participants who complete the study. The intervention will be considered feasible if no more than 20% of participants are lost to follow up.
Time Frame: 3 months post randomization
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention | Usual Care
Number analyzed (Participants) | 7 | 7 | 0
Participants | 7 | 7 | 0

2. Primary Outcome: Percentage of Participants That Are Enrolled and Attend the Study the Study Sessions Compared to Enrolled
Description: Acceptability of the intervention will be operationalized as study session attendance and will be considered adequate if at least 70% of the sessions are attended.
Time Frame: 3 months post randomization
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention | Usual Care
Number analyzed (Participants) | 7 | 7 | 0
Participants | 7 | 7 | 0

3. Secondary Outcome: Change in Hemoglobin A1c (HbA1C) Level
Description: Hemoglobin A1c (HbA1C) in % will be measured via blood draw and processing. Normal values HbA1C are less than 5.7%, values between 5.7% and 6.4% indicate pre-diabetes, and persons with levels of 6.5% or higher are considered to have diabetes.
Time Frame: Baseline and 3 months post randomization
Population: The A1C results may be affected by variations in point of care vs regular blood testing and the timing of follow up for participants. Data is included for participants who completed more than 65% of the intervention sessions.
Measure: Mean (Standard Deviation); unit: percentage of HbA1C
Groups:
- Group-based Cognitive Behavioral Intervention: Subjects receiving the group-based CT-CBintervention Group-based CognitiveBehavioral Intervention: This intervention will include six 1-hour group sessions held biweekly for twelve weeks. Each sixty-minute session will consist of 15 minutes of diabetes education regarding exercise and food planning and approximately 45 minutes of CT-CB presentations/engagement activities. Participants will be encouraged to bring along their family members or friends for support.
- Web-based Cognitive Behavioral Intervention: Subjects receiving the web-based CT-CBintervention Web-based CognitiveBehavioralIntervention: This intervention will include six 1-hour web-based sessions held biweekly for twelve weeks. Subjects in the web-based CT-CB will be asked to reserve a 1hour period for a web call from the behavioral interventionist team. Text reminders will be sent to the participants prior to the sessions. During this period, approximately 15minutes will be reserved for diabetes exercise and food planning education and approximately 45minutes of CT-CBengagement activities.
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention
Number analyzed (Participants) | 7 | 7
percentage of HbA1C
  Baseline | 10.35 (1.01) | 9.67 (1.39)
  Month 3 | 9.21 (0.91) | 8.74 (2.06)

4. Secondary Outcome: Change in Patient Health Questionnaire (PHQ-9) Score
Description: Depressive symptoms are assessed by the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a 9-item scale where respondents indicate how much they are bothered by certain problems on a 4-point scale where 0 = not at all and 3 = nearly every day. Total scores range from 0 to 27 with degree of depression considered minimal for scores between 0-4, mild for scores of 5-9, moderate for scores of 10-14, moderate to severe for scores 15-19, and severe for scores of 20-27.
Time Frame: Baseline and 3 months post randomization
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention | Usual Care
Number analyzed (Participants) | 7 | 7 | 0
Score on a scale
  Baseline | 7.29 (5.47) | 6.00 (4.90) |
  3 months post randomization | 7.71 (6.92) | 5.00 (3.87) |

5. Secondary Outcome: Change in Diabetes Distress Scale (DDS17) Score
Description: The Diabetes Distress Scale (DDS17) is a 17-item questionnaire assessing the severity of problems of living with diabetes. Participants indicate the degree to which each item impacts their life on a 6-point scale where 1 = not a problem and 6 = a very serious problem. The scores are summed and divided by 17 to generate an average score that can range from 1 to 6. Scores of 3 or more are considered high distress.
Time Frame: Baseline and 3 months post randomization
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention | Usual Care
Number analyzed (Participants) | 7 | 7 | 0
score on a scale
  Baseline | 2.35 (0.82) | 2.57 (0.90) |
  3 months post randomization | 1.74 (0.64) | 2.15 (0.99) |

6. Secondary Outcome: Change in 12-Item Short Form Health Survey (SF-12) Score
Description: Quality of life will be assessed with the 12-Item Short Form Health Survey (SF-12). The Short Form-12 Health Survey Questionnaire (SF-12) is a measure of general physical and mental health. The SF-12 consists of 12 items with a Likert-type response format that measures quality of life with a Physical Component Summary (PCS) and Mental Component Summary (MCS). Subscales associated with the PCS include physical functioning, role limitations due to physical problems, bodily pain, and general health perceptions. Subscales associated with the MCS include vitality (energy and fatigue), social functioning, role limitations due to emotional problems, and mental health. A scoring algorithm is used to generate a total score for each component ranging from 0 to 100. Low values represent a poor health state while high values represent a good health state.
Time Frame: Baseline and 3 months post randomization
Population: There was an error in data collection forms provided to participants, which made these questionnaires unusable for data analysis.
Groups:
- Group-based or Web-based Cognitive Behavioral Intervention: Participants from both study arms are combined for this analysis.
Arm/Group | Group-based or Web-based Cognitive Behavioral Intervention
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Generalized Anxiety Disorder 7-item (GAD-7) Scale Score
Description: Anxiety will be assessed using the Generalized Anxiety Disorder 7-item (GAD-7) Scale. Participants use a 4-point scale in response to statements about anxiety (such as "trouble relaxing") to indicate how bothered they have felt by item over the last two weeks. Degree of anxiety is rated as 0 = "not at all" to 3 = "nearly every day". Total scores range from 0 to 21. Scores of 5-9 indicate mild anxiety, 10-15 indicates moderate anxiety and scores 15 and greater indicate severe anxiety.
Time Frame: Baseline and 3 months post randomization
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention | Usual Care
Number analyzed (Participants) | 7 | 7 | 0
score on a scale
  Baseline | 7.14 (4.63) | 5.57 (7.28) |
  3 months post randomization | 6.00 (5.80) | 2.43 (4.47) |

8. Secondary Outcome: Change in Self Efficacy for Diabetes
Description: Change in Self Efficacy is assessed by Self Efficacy for Diabetes Scale that is administered at Baseline and at 3rd month post randomization. The questionnaire is a 8 item scale. Each question ranks from 1(not confident at all) to 10 (totally confident). The scale score will be compared from Baseline to 3 months post randomization.
  For diabetes, higher diabetes self-efficacy has been shown to relate to better self-care and glycaemic control. Increase in the score of Self-efficacy is found to directly reinforce adherence to self-care.
Time Frame: Baseline and 3 months post randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Web-based Cognitive Behavioral Intervention: Subjects receiving the web-based CT-CB intervention
  Web-based Cognitive Behavioral Intervention: This intervention will include six 1-hour web-based sessions held biweekly for twelve weeks. Subjects in the web-based CT-CB will be asked to reserve a 1 hour period for a web call from the Behavioral Interventionist team. Text reminders will be sent to the participants prior to the sessions. During this period, approximately 15 minutes will be reserved for diabetes exercise and food planning education and approximately 45 minutes of CT-CB engagement activities.
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention
Number analyzed (Participants) | 7 | 7
score on a scale
  Baseline | 7.34 (1.43) | 6.94 (2.10)
  3 months post randomization | 7.43 (2.20) | 6.77 (1.84)

9. Secondary Outcome: Change in Diabetes Health Belief Scale
Description: Change in Diabetes Health Belief Scale is assessed by 25-item scale that is administered at baseline and at 3 months post randomization.Each question ranks from (1 = Strongly Disagree) to (5 = Strongly Agree).The scale score will be compared from Baseline to 3 months post randomization
Time Frame: Baseline and 3 months post randomization
Population: This survey was not administered to participants.
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention | Usual Care
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Three months post-randomization
Description: Adverse events such as episodes of hypoglycemia, diabetes-related hospitalizations, and ER or urgent care visits will be ascertained during the study visits.
Arm/Group | Group-based Cognitive Behavioral Intervention | Web-based Cognitive Behavioral Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/0
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated. A control group was intended to be added for the study, but the study team decided not to complete this additional research due to the COVID pandemic. Additional funds were not available to enroll the control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03562767/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT03562767/ICF_001.pdf